CLINICAL TRIAL: NCT06679543
Title: Effects of Partial Sleep Deprivation on Cardiac Output During Cycling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Philip Millar, Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24-03-017
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep Deprivation
Keywords: exercise blood pressure; cardiac output; plasma volume; sleep deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep (No Intervention): During this arm, participants will be asked to come to the lab for testing after a night of normal sleep. Normal sleep will be defined as participants habitual sleep-wake timing.
- Partial sleep deprivation (Experimental): During this arm, participants will be asked to come to the lab for testing after a night of partial sleep deprivation. Participants will be asked to fall asleep at their habitual bedtime but wake up early (~40% of normal sleep duration).
  Interventions: Other: Partial sleep deprivation

INTERVENTIONS:
Other: Partial sleep deprivation — Participants will be asked to come to the lab for testing after a night of partial sleep deprivation. Participants will be asked to fall asleep at their habitual bedtime but wake up early (~40% of normal sleep duration).
  Arms: Partial sleep deprivation

SUMMARY:
The goal of this clinical trial is to determine if attenuations in cardiac output drive the blunted blood pressure response during cycling exercise following a night of partial sleep deprivation in young healthy adults (%50 females). The secondary outcome is to assess sex differences. The main questions it aims to answer are:

* Do reductions in plasma volume drive reductions in cardiac output and therefore blood pressure during exercise following a night of partial sleep deprivation?
* Do sex differences exist?

Participants will:

* Visit the lab after a night of normal sleep and a night of partial sleep deprivation.
* Keep a daily diary of their sleep and food/beverage intake.
* Perform maximal and submaximal exercise on a cycle ergometer.

DETAILED DESCRIPTION:
The investigators recently published data showing systolic blood pressure is attenuated during cycling exercise in males but not females following acute partial sleep deprivation, compared to a night of normal sleep, despite no differences in power output. The mechanisms responsible for this sex difference remain unknown. The investigators have pilot data that suggests males have a reduction in cardiac output following acute partial sleep deprivation, but females do not. Therefore, the primary purpose of this study is to assess hemodynamics (blood pressure, stroke volume, and cardiac output) and plasma volume during cycling exercise following a night of normal sleep and partial sleep deprivation in otherwise healthy males and females.

Thirty young healthy adults (50% female) will be recruited to undergo three visits. The first visit will assess maximal oxygen uptake to determine aerobic fitness and metabolic exercise intensity zones. The following two testing visits will be randomized and will be completed after a night of normal sleep or acute partial sleep deprivation (early awakening, 40% normal sleep duration). Sleep will be measured 1-week before each visit subjectively (questionnaire) to determine habitual sleep timing and duration and objectively (wrist actigraphy) the night before each testing visit. Each testing visit will require participants to complete a constant load 60-minute bout of cycling. Before, during, and after the exercise protocol, the investigators will measure hemodynamics and plasma volume. Venous blood samples will be collected via intravenous lines.

ELIGIBILITY:
Inclusion Criteria:

* Free of known cardiovascular or metabolic diseases or sleep disorders
* No history of smoking (within the past 3 months)
* Able to engage in physical activity assessed through the physical activity readiness questionnaire (PAR-Q+)
* No prescription of chronic medications other than oral contraceptives
* Able to abide by sleep protocols for all visits
* Individuals who are not allergic to ultrasound gel
* Individuals who are not pregnant

Exclusion Criteria:

* Individuals diagnosed with cardiovascular or metabolic disease or sleep disorders
* Has a history of smoking (within the past 3 months)
* Not ready to engage in physical activity as assessed by the PAR-Q+
* Individuals prescribed chronic medications other than oral contraceptives
* Unable to abide by sleep protocols for any testing visit
* Allergic to ultrasound gel
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
cardiac output responses to cycling exercise | Comparison between normal sleep and partial sleep deprivation, ~3 weeks
  Cardiac output during exercise after a night of normal sleep and after a night of partial sleep deprivation

SECONDARY OUTCOMES:
Blood pressure responses to cycling exercise | Comparison between normal sleep and partial sleep deprivation, ~3 weeks
  Blood pressure during exercise after a night of normal sleep and after a night of partial sleep deprivation
Plasma volume | Comparison between normal sleep and partial sleep deprivation, ~3 weeks
  Plasma volume after a night of normal sleep and after a night of partial sleep deprivation

CONTACTS AND LOCATIONS:
Overall Officials: Julian Bommarito, MSc, Study Director — University of Guelph; Philip Millar, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Time Frame: Beginning after publication with no end date